CLINICAL TRIAL: NCT05089916
Title: Radiation During Osimertinib Treatment: a Safety and Efficacy Cohort Study
Acronym: ROSE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-YMO/TRK-0120; 2022-503028-29-01 (EU CTIS Number); 2020-003512-27 (EudraCT Number)
Record Dates: First submitted 2021-04-13; First posted 2021-10-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: NSCLC; EGFR Positive Non-small Cell Lung Cancer; Oligoprogression
Keywords: Osimertinib; Radiotherapy; TKI
MeSH Terms: interventions — osimertinib; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Single arm, explorative, multi-center parallel cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib plus Radiation (Experimental): Osimertinib 80 mg Radiation as per SOC
  Interventions: Drug: Osimertinib; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Osimertinib — Osimertinib: according to its marketing authorization, i.e. at daily doses of 80 mg, for a maximum of 12 months within the study.
  Other Names: Tagrisso
Radiation: Radiotherapy — Radiotherapy: according to standard of care
  The target population will comprise 3 parallel cohorts, for cohort 1 and 3 a minimum of 10 subjects is planned to be enrolled:
  1. Irradiation of bone, solid organ (non-lung, non-brain) or soft-tissue metastases
  2. Irradiation of brain metastases (initial lesion size < 3 cm)
  3. Irradiation of lung lesions (primary tumor or metastases, lesion size < 5 cm)

SUMMARY:
Study Objectives are:

To assess the safety of osimertinib treatment continuation during irradiation therapy for palliation or oligoprogressive disease by assessment of grade 3-5 AEs during and after concomitant osimertinib and irradiation of tumor sites.

To assess the efficacy of osimertinib treatment continuation during irradiation therapy for palliation or oligoprogressive disease.

To investigate Quality of Life during and after irradiation therapy and concomitant osimertinib.

DETAILED DESCRIPTION:
Many patients with advanced lung cancer require palliative irradiation of metastases to relieve symptoms and prevent local complications. In addition, guidelines recommend local treatment (including radiation) for oligoprogression during TKI treatment. Clinicians are faced with the decision whether to continue TKI therapy during irradiation, a practice for which there is little data, or to interrupt the oral treatment for the duration of radiation, which may lead to progression of non-irradiated lesions. For erlotinib and gefitinib there is some data indicating that cranial irradiation as well as stereotactic body irradiation may be carried out safely without discontinuing or interrupting the TKI treatment. Although some small case series report on a PFS benefit with irradiation during osimertinib treatment, there is very limited data on the safety of osimertinib during irradiation, and no evidence-based recommendations around stopping osimertinib for irradiation.

The hypothesis is that osimertinib can be continued without interruption during irradiation of individual tumor lesions in the setting of oligoprogressive NSCLC, or for local symptom control of primary tumor or metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study specific procedures, including screening evaluations that are not SOC.
2. Age ≥ 18 years at time of study entry.
3. Histologically confirmed NSCLC
4. Ongoing or planned osimertinib treatment according to marketing authorization (first line treatment of tumor positive for a common or uncommon EGFR mutation, or later line treatment of tumor positive for EGFR T790M mutation, assessed according to local standard. First line therapy is defined as therapy used to treat advanced disease. Each subsequent line of therapy is preceded by disease progression. A switch of an agent within a regimen in order to manage toxicity does not define the start of a new line of therapy. Experimental therapies when given as separate regimen are considered as separate line of therapy. Maintenance therapy following platinum doublet-based chemotherapy is not considered as a separate regimen of therapy.)
5. Clinical indication for radiotherapy of one or more lesions, for instance for local symptom control of primary tumor or metastasis, for oligoprogressive metastasis, or for disease control with conventional or stereotactic strategy. Radiotherapy of metastatic sites can be for bone, solid organ or soft-tissue lesions; initial size of brain metastases should be < 3 cm. Lung lesions should be no more than 5 cm.
6. ECOG performance status 0-2.
7. Life expectancy ≥12 weeks
8. Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged 50 years or more and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution.
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
9. Male subjects who are sexually active with WOCBP should be willing to use highly effective contraception. Men who are azoospermic do not require contraception.
10. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
11. Negative COVID-19 test within 1 week prior to starting irradiation if clinically required by current regional COVID-19 outbreak situation.

Exclusion Criteria:

1. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study, or during the follow-up period of an interventional study.
2. Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater
3. Previous enrolment in the present study.
4. Any chemotherapy, biologic or hormonal cancer therapy other than EGFR-TKIs used concurrently or within 4 weeks prior to study enrolment, or checkpoint inhibitors within 130 days prior to study enrolment. Hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
5. Any unresolved toxicities from prior therapy greater than grade I (exception: alopecia, grade 2 neuropathy) which in the investigator's opinion would jeopardise compliance with the protocol or worsen during irradiation
6. Cardiac side-effects of osimertinib not sufficiently improved by dose reduction as suggested by the label/ German "Fachinformation".
7. In patients with indication for radiotherapy of lung lesions: past medical history of ILD/pneumonitis, radiation pneumonitis grade 2 or higher (CTCAE V5.0) or requiring steroid treatment, or any evidence of clinically active ILD, in particular interstitial pulmonary fibrosis (IPF).
8. Major surgery (as defined by the Investigator) within 4 weeks prior to starting the study; patients must have recovered from effects of preceding major surgery. Note: Local non-major surgery for palliative intent (e.g., surgery of isolated lesions) is acceptable.
9. Congenital long QT syndrome
10. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value
    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block.
    * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN) , congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes
11. Inadequate bone marrow reserve or organ function (as demonstrated by any of the following laboratory values:

    * Absolute neutrophil count <1.5 x 109/L;
    * Platelet count <100 x 109/L;
    * Hemoglobin <90 g/L (9 g/dL);
    * Alanine aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
    * Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
    * Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinemia] or liver metastases;
    * Serum creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min [measured or calculated by Cockcroft and Gault equation]-confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
12. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection.
13. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
14. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
15. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
16. Active infection will include any patients receiving treatment for infection.
17. Clinical suspicion of COVID-19 with or without negative COVID-19 test
18. Participants with HBV infection are eligible only if they meet the following criteria:

    * Demonstrated absence of HCV co-infection or history of HCV co-infection
    * Demonstrated absence of HIV infection
    * Participants with active HBV infection are eligible if:
    * they are receiving anti-viral treatment for at least 6 weeks prior to study treatment,
    * HBV DNA is suppressed to <100 IU/mL,
    * transaminase levels are below ULN.

    Participants with a resolved or chronic HBV infection are eligible if they are:

    • Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc IgG] In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment.

    or

    • Positive for HBsAg, but for > 6 months have had transaminases levels below ULN and HBV DNA levels <100 IU/mL (i.e., are in an inactive carrier state). In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment. Refer to section "5.5.2. Special warnings and precautions"

    Participants with HIV infection are only eligible if they meet all the following criteria:
    * Undetectable viral RNA load for 6 months
    * CD4+ count of >350 cells/μL
    * No history of AIDS-defining opportunistic infection within the past 12 months
    * Stable for at least 4 weeks on the same anti-HIV medications
19. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
20. Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 week prior). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
21. Women who are pregnant or breast-feeding
22. Male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 4 months after the last dose of osimertinib
23. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Frequency, time of onset and severity of Adverse Events as assessed by investigator during osimertinib treatment and irradiation therapy | 24 months
  Safety and tolerability (Frequency, time of onset and severity of Adverse Events, grading according to CTCAE V5.0), including pneumonitis, interstitial lung disease, radiation pneumonitis, radionecrosis, radiation alveolitis, radiation fibrosis - lung, pulmonary radiation injury and cardiac failure (congestive heart failure - CHF) as adverse events of special interest

SECONDARY OUTCOMES:
PFS | 24 months
  Progression-free survival: calculated as PFS1, PFS2, PFS3, PFS0 to assess osimertinib treatment continued beyond several progression events entailing radiotherapy, and prior to first radiotherapy
TTF | 12 months
  Time to treatment failure
Local tumor control | 24 months
  Local tumor control
OS | 24 months
  Overall survival
QoL | 12 months
  Quality of Life assessed by EORTC QLQ-C30

OTHER OUTCOMES:
Blood sample analysis and biomarker assessment | 24 months
  To explore blood-based biomarkers in this setting
Tissue-based biomarkers | Before or within 3 weeks after start of study treatment
  Optional tumor tissue analysis (pre-study FFPE sample) and biomarker correlation with patient baseline characteristics and outcomes
Target volume of irradiation | 28 days
  To investigate target volumes used.
Type of irradiation | 28 days
  To investigate types of irradiation (conventional vs. stereotactic)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Tufman, Prof. Dr., Principal Investigator — LMU Klinikum der Universität München
Locations (1):
- LMU Klinikum der Universität München, München, Germany

IPD SHARING:
Plan to Share IPD: No